CLINICAL TRIAL: NCT07185464
Title: Efficacy and Safety of Transcranial Alternating Current Stimulation (tACS) in Adolescents With First-episode Depression Who Are Drug-naive: A Randomized, Double-blind, Controlled Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1stChongqingMU___ZXY
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This study adopts a parallel assignment design. Participants will be randomized in a 1:1 ratio to either the active tACS group or the sham stimulation group, with all participants receiving oral sertraline throughout the trial. The intervention group will undergo 20 sessions of active tACS over 4 weeks, while the control group will receive sham stimulation using an identical device that delivers no current. Participants will remain in their assigned group for the entire duration of the study without crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tACS (Experimental): Participants in this group will receive transcranial alternating current stimulation (tACS) in addition to daily oral sertraline. tACS will be administered using the NEXALIN ADI device (Beijing Neslin Technology Co., Ltd.) with stimulation parameters set at a frequency of 77.5 Hz and a current intensity of 15 mA. One electrode will be placed on the forehead and two electrodes on the mastoid processes. Each session will last approximately 40 minutes, with a total of 20 sessions delivered across 4 consecutive weeks (5 sessions per week). The intervention is designed to modulate abnormal cortical oscillations, thereby alleviating depressive symptoms, enhancing cognitive performance, and supporting emotional regulation.
  Interventions: Device: tACS
- Sham (Sham Comparator): Arm Description: Participants in this group will receive sham stimulation in addition to daily oral sertraline. A sham device, identical in appearance, sound, and operation to the active tACS device, will be used but will not deliver any electrical current. Sessions will follow the same schedule as the active group (20 sessions over 4 weeks, 5 sessions per week). Both participants and operators will remain blinded to treatment allocation to maintain trial integrity.
  Interventions: Device: tACS

INTERVENTIONS:
Device: tACS — This intervention uses the NEXALIN ADI alternating current stimulation device from Beijing Naisilin Technology Co., Ltd., to deliver targeted stimulation to the prefrontal cortex and bilateral mastoid regions. The prefrontal cortex electrode directly stimulates the cerebral cortex, while the mastoid electrodes ensure the synchronized activation of bilateral neural pathways. Stimulation is applied at a frequency of 77.5 Hz and a current intensity of 15 mA, aiming to optimize brainwave synchronization and modulate brain activity. Participants will undergo daily sessions lasting approximately 40 minutes each, for a total of 20 sessions over 4 weeks. The non-invasive nature of the intervention, combined with its precise targeting of specific brain regions, distinguishes it from other neuromodulation therapies. The treatment aims to enhance neural synchronization, promote neuroplasticity, and provide a non-pharmacological therapeutic alternative for patients.
  Arms: tACS
Device: tACS — In the sham stimulation group, participants will receive intervention using a sham device that is identical in appearance, operation, and stimulation protocol to the real tACS device, but does not deliver any current. Both participants and operators will be unable to distinguish between real and sham stimulation based on the device's appearance, sound, or tactile feedback. Device allocation will follow a randomized code generated in advance to ensure blinding and proper group assignment.
  Arms: Sham

SUMMARY:
To evaluate the efficacy of tACS treatment.To determine whether tACS can accelerate symptom remission, improve clinical response rates, and facilitate the recovery of emotional and cognitive functions through standardized clinical assessments.To evaluate the safety of tACS treatment.To assess adverse events and side effects in both the intervention and control groups, ensuring the safety and tolerability of tACS in adolescent populations.

DETAILED DESCRIPTION:
This randomized, double-blind, sham-controlled pilot trial will evaluate the efficacy and safety of transcranial alternating current stimulation (tACS) combined with sertraline in adolescents with first-episode, drug-naive major depressive disorder (MDD). Eligible participants are aged 12-18 years, meet DSM-5 criteria for a current depressive episode confirmed by K-SADS-PL, have a CDRS-R score ≥40, and have not received antidepressant treatment during the current episode.A total of 30 participants will be randomized 1:1 to receive either active tACS or sham stimulation, in addition to oral sertraline (25 mg/day in the first week, titrated to 50 mg/day thereafter). The active group will undergo 20 sessions over 4 weeks (5 sessions per week) using the NEXALIN ADI device (77.5 Hz, 15 mA, 40 minutes per session). The sham device is identical in appearance but delivers no current. Both participants and operators will remain blinded.Primary outcomes are changes in depressive symptoms, measured by the CDRS-R and BDI. Secondary outcomes include anxiety (SCARED, HAMA), global improvement (CGI-S, CGI-I), mania symptoms (YMRS), suicide risk (C-SSRS), quality of life (PedsQL4.0), sleep (PSQI), rumination (RSS), and cognition (THINC-it). Safety will be monitored through adverse events, vital signs, laboratory tests, and tolerability assessments.This pilot study will provide preliminary evidence on the potential of tACS as an adjunctive treatment for adolescent depression and inform future large-scale trials.

ELIGIBILITY:
Inclusion Criteria:

1.Age 12-18 years; 2.Subjects met the diagnostic criteria for depression in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) as determined by the Childhood Affective Disorders and Schizophrenia Questionnaire (K-SADS-PL) and were currently in a depressive episode; 3.Children's Depression Rating Scale-Revised (CDRS-R) score ≥ 40 points; 4.Not receiving any antidepressant medication during the current depressive episode.

Exclusion Criteria:

1.Other comorbid mental disorders in accordance with DSM-5 except anxiety disorders; 2.Depression with psychotic symptoms; 3.Young Mania Rating Scale (YMRS) > 13; 4.History of neurological disease (such as epilepsy, brain trauma, etc.) or serious physical disease (such as thyroid disease, lupus erythematosus, diabetes, lung, liver and kidney damage, major trauma, etc.); 5.Previous treatment with electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), tACS or other neurostimulation treatments; 6.Patients currently receiving anti-epileptic drugs or high-dose benzodiazepines; 7.History of alcohol or drug abuse or dependence; 8.Breastfeeding women or pregnant women; 9.Contraindications to MRI; 10.Currently at high risk of suicide.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in CDRS-R (Children's Depression Rating Scale) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  Clinical response (≥ 50% reduction in CDRS-R scores from baseline)

SECONDARY OUTCOMES:
Change in BDI-II (Baker Depression Scale) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  Change in BDI-II (Baker Depression Scale) scores from baseline
Change in SCARED (The Screen for Child Anxiety-Related Emotional Disorders) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  Improvement in anxiety (SCARED minus the scores）
Change in suicide risk from baseline on the C-SSRS (Columbia Suicide Severity Rating Scale) | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  The severity of the suicide risk
Change in PSQI (Pittsburgh Sleep Quality Index) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  Improvement in sleep status (PSQI minus the scores）
Change in PedsQL4.0 (The Pediatric Quality of Life Inventory) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  Improvement of children's quality of life（PedsQL4.0 minus the scores)
Change in CGI-S (Clinical Global Impressions-Severity Scales) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  Improvement in overall clinical impression severity ( 7-point scale, with 1 being normal and 7 being among the most severely damaged )
Change in CGI-I (Clinical Global Impressions-Improvement Scales) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  Improvement of clinical general Impression scale (7-point scale,7 denoting a very significant deterioration)
Change in RSS (Ruminative Responses Scale) | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months.
  The level of improvement in negative thinking(the higher the total score, the more reflective thinking the more severe it is).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Hetrick SE, McKenzie JE, Bailey AP, Sharma V, Moller CI, Badcock PB, Cox GR, Merry SN, Meader N. New generation antidepressants for depression in children and adolescents: a network meta-analysis. Cochrane Database Syst Rev. 2021 May 24;5(5):CD013674. doi: 10.1002/14651858.CD013674.pub2. PMID 34029378
- [Background] Clancy KJ, Andrzejewski JA, You Y, Rosenberg JT, Ding M, Li W. Transcranial stimulation of alpha oscillations up-regulates the default mode network. Proc Natl Acad Sci U S A. 2022 Jan 4;119(1):e2110868119. doi: 10.1073/pnas.2110868119. PMID 34969856
- [Background] Jones KT, Johnson EL, Gazzaley A, Zanto TP. Structural and functional network mechanisms of rescuing cognitive control in aging. Neuroimage. 2022 Nov 15;262:119547. doi: 10.1016/j.neuroimage.2022.119547. Epub 2022 Aug 5. PMID 35940423
- [Background] Yan CG, Chen X, Li L, Castellanos FX, Bai TJ, Bo QJ, Cao J, Chen GM, Chen NX, Chen W, Cheng C, Cheng YQ, Cui XL, Duan J, Fang YR, Gong QY, Guo WB, Hou ZH, Hu L, Kuang L, Li F, Li KM, Li T, Liu YS, Liu ZN, Long YC, Luo QH, Meng HQ, Peng DH, Qiu HT, Qiu J, Shen YD, Shi YS, Wang CY, Wang F, Wang K, Wang L, Wang X, Wang Y, Wu XP, Wu XR, Xie CM, Xie GR, Xie HY, Xie P, Xu XF, Yang H, Yang J, Yao JS, Yao SQ, Yin YY, Yuan YG, Zhang AX, Zhang H, Zhang KR, Zhang L, Zhang ZJ, Zhou RB, Zhou YT, Zhu JJ, Zou CJ, Si TM, Zuo XN, Zhao JP, Zang YF. Reduced default mode network functional connectivity in patients with recurrent major depressive disorder. Proc Natl Acad Sci U S A. 2019 Apr 30;116(18):9078-9083. doi: 10.1073/pnas.1900390116. Epub 2019 Apr 12. PMID 30979801
- [Background] Chai Y, Gehrman P, Yu M, Mao T, Deng Y, Rao J, Shi H, Quan P, Xu J, Zhang X, Lei H, Fang Z, Xu S, Boland E, Goldschmied JR, Barilla H, Goel N, Basner M, Thase ME, Sheline YI, Dinges DF, Detre JA, Zhang X, Rao H. Enhanced amygdala-cingulate connectivity associates with better mood in both healthy and depressive individuals after sleep deprivation. Proc Natl Acad Sci U S A. 2023 Jun 27;120(26):e2214505120. doi: 10.1073/pnas.2214505120. Epub 2023 Jun 20. PMID 37339227
- [Background] Wang J, Zhao W, Wang H, Leng H, Xue Q, Peng M, Min B, Jin X, Tan L, Gao K, Wang H. Brain-wide activation involved in 15 mA transcranial alternating current stimulation in patients with first-episode major depressive disorder. Gen Psychiatr. 2024 Mar 8;37(2):e101338. doi: 10.1136/gpsych-2023-101338. eCollection 2024. PMID 38476648
- [Background] Biackova N, Adamova A, Klirova M. Transcranial alternating current stimulation in affecting cognitive impairment in psychiatric disorders: a review. Eur Arch Psychiatry Clin Neurosci. 2024 Jun;274(4):803-826. doi: 10.1007/s00406-023-01687-7. Epub 2023 Sep 8. PMID 37682331
- [Background] Zhou J, Li D, Ye F, Liu R, Feng Y, Feng Z, Li R, Li X, Liu J, Zhang X, Zhou J, Wang G. Effect of add-on transcranial alternating current stimulation (tACS) in major depressive disorder: A randomized controlled trial. Brain Stimul. 2024 Jul-Aug;17(4):760-768. doi: 10.1016/j.brs.2024.06.004. Epub 2024 Jun 14. PMID 38880208
- [Background] Elyamany O, Leicht G, Herrmann CS, Mulert C. Transcranial alternating current stimulation (tACS): from basic mechanisms towards first applications in psychiatry. Eur Arch Psychiatry Clin Neurosci. 2021 Feb;271(1):135-156. doi: 10.1007/s00406-020-01209-9. Epub 2020 Nov 19. PMID 33211157
- [Background] Bowes L, Joinson C, Wolke D, Lewis G. Peer victimisation during adolescence and its impact on depression in early adulthood: prospective cohort study in the United Kingdom. Br J Sports Med. 2016 Feb;50(3):176-83. doi: 10.1136/bjsports-2015-h2469rep. PMID 26782765
- [Background] Consoli A, Peyre H, Speranza M, Hassler C, Falissard B, Touchette E, Cohen D, Moro MR, Revah-Levy A. Suicidal behaviors in depressed adolescents: role of perceived relationships in the family. Child Adolesc Psychiatry Ment Health. 2013 Mar 16;7(1):8. doi: 10.1186/1753-2000-7-8. PMID 23497551
- [Background] Hankin BL. Depression from childhood through adolescence: Risk mechanisms across multiple systems and levels of analysis. Curr Opin Psychol. 2015 Aug;4:13-20. doi: 10.1016/j.copsyc.2015.01.003. PMID 25692174
- [Background] Barker MM, Beresford B, Bland M, Fraser LK. Prevalence and Incidence of Anxiety and Depression Among Children, Adolescents, and Young Adults With Life-Limiting Conditions: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Sep 1;173(9):835-844. doi: 10.1001/jamapediatrics.2019.1712. PMID 31282938
- [Background] Beardslee WR, Brent DA, Weersing VR, Clarke GN, Porta G, Hollon SD, Gladstone TR, Gallop R, Lynch FL, Iyengar S, DeBar L, Garber J. Prevention of depression in at-risk adolescents: longer-term effects. JAMA Psychiatry. 2013 Nov;70(11):1161-70. doi: 10.1001/jamapsychiatry.2013.295. PMID 24005242